CLINICAL TRIAL: NCT06217120
Title: Reversing Microvascular Dysfunction in Heart Failure With Ejection Fraction > 40% Using Colchicine (The COL-Micro-HF Study)
Brief Title: Reversing Microvascular Dysfunction in Heart Failure With Preserved Ejection Fraction
Acronym: COL-Micro-HF
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICM 2024-3370
Record Dates: First submitted 2023-11-29; First posted 2024-01-22 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Microvascular Coronary Artery Disease
Keywords: Heart Failure with Preserved Ejection Fraction; Microvascular Coronary Artery Disease; Inflammation; Colchicine
MeSH Terms: conditions — Inflammation | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: This will be a pilot mechanistic study. Patients will be randomly assigned in a 1:1 ratio to receive colchicine 0.5 mg daily or a matched placebo. Follow-up will occur at 6 months after randomization.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COLCHICINE (Active Comparator)
  Interventions: Drug: Colchicine
- PLACEBO (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine — Colchicine 0.5 mg daily
  Arms: COLCHICINE
Drug: Placebo — Placebo once daily
  Arms: PLACEBO

SUMMARY:
This study will evaluate the impact of colchicine on the change in coronary flow reserve (CFR), a marker for coronary microvascular dysfunction (CMD), compared to placebo in patients with heart failure and ejection fraction above 40% (including patients with improved EF).

DETAILED DESCRIPTION:
This will be a pilot mechanistic study. Patients will be randomly assigned in a 1:1 ratio to receive colchicine 0.5 milligram (mg) daily or a matched placebo. Follow-up will occur six months after randomization.

The study aims to test the impact of reducing inflammation using a pharmacological strategy to reverse CMD in patients with HF and EF above 40%. The investigators will test the effect of colchicine on the change in coronary flow reserve (CFR), a marker for CMD, compared to placebo. The investigators will assess CMD using adenosine-based positron emission tomography (PET).

The primary objective will be to compare changes in CFR between six months and baseline according to therapy.

The primary Endpoint will be the change from baseline to 6 months in CFR, a marker of CMD.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 40 years of age,
2. Chronic symptomatic HF and left ventricular ejection fraction (LVEF) > 40% within 12 months prior to the screening visit (regardless of the imaging modality) documented by one of the following:

   1. HF requiring hospitalization and IV diuretics within 12 months of study entry, or
   2. NTproBNP > or = 150pg/ml in sinus rhythm or NTproBNP > or = 450pg/ml in chronic atrial fibrillation,
3. New York Heart Association Class, NYHA functional class II to (ambulatory) IV,
4. Evidence of pathological systemic inflammation: high C-reactive protein, hs-CRP levels (hs-CRP > or = 5mg/L),
5. Subjects with the capacity to provide informed consent.

Exclusion Criteria:

1. Patients with a diagnosis of infiltrative cardiomyopathy,
2. Presence of severe valvular heart disease,
3. Presence of active infection within the 3 months prior to enrollment needing antibiotics (excluding COVID (Coronavirus disease)-19),
4. Acute decompensated HF, acute coronary syndrome (including MI), cardiac surgery, other major cardiovascular surgery, or urgent percutaneous coronary intervention (PCI) within the 3 months prior to enrollment,
5. Known or clinically judged significant (i.e., angina with CCS (Canadian Cardiovascular Society) class > 2/4) epicardial coronary artery disease (CAD) that has not been revascularized (revascularized CAD is defined by a history of myocardial infarction, percutaneous intervention, or coronary artery bypass grafting),
6. History of hypersensitivity to colchicine,
7. Evidence of hepatic disease as determined by any 1 of the following: AST or ALT values exceeding 3× the upper limit of normal at enrollment; or patient with a history of cirrhosis, chronic active hepatitis, or severe hepatic disease,
8. Patients with estimated glomerular filtration rate (eGFR) <30 ml/min/1.73 m2 as calculated by the Modification in Diet in Renal Disease (MDRD) formula at enrollment,
9. Subject with inflammatory bowel disease (Crohn's disease or ulcerative colitis) or patient with chronic diarrhea,
10. Patient with pre-existent progressive neuromuscular disease,
11. Patient currently taking colchicine for other indications (mainly chronic indications represented by Familial Mediterranean Fever or gout). There is no wash-out period required for patients who have been treated with colchicine and stopped treatment prior to enrolment,
12. Patients under long-term steroid medication for a chronic condition,
13. Contraindication to dipyridamole-containing medication, acute myocardial infarction or unstable angina in the past 48h,
14. Positive pregnancy test results at the screening visit, and females of childbearing potential who do not agree to use adequate methods of contraception for the duration of the study; acceptable means of birth control include: implantable contraceptives, injectable contraceptives, oral contraceptives, transdermal contraceptives, intrauterine devices, male or female condoms with spermicide, abstinence, or a sterile sexual partner,
15. History or presence of any other disease with a life expectancy of <1 year,
16. Patient considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in coronary flow reserve (CFR) between baseline and six months | Baseline and 6 months
  The primary endpoint will be the change from baseline to 6 months in CFR, a marker of coronary microvascular dysfunction (CMD), according to therapy (colchicine vs. placebo). Assessment of CFR will be based on 82-Rubidium Positron emission tomography (82Rb-PET)-myocardial perfusion imaging, performed at baseline and 6-month follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol